CLINICAL TRIAL: NCT02286986
Title: A 2-part Study to Investigate the Dose-ranging Pharmacokinetics and Tolerability, Followed by the Efficacy and Safety of Cannabidiol (GWP42003-P) in Children and Young Adults With
Brief Title: Cannabidiol (CBD) to 27 Patients (Aged 2 Years - 19 Years) With Drug Resistant Epilepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Francis Filloux, Francis M. Filloux, M.D. Division Chief, Pediatric Neurology University of Utah School of Medicine, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 70871
Record Dates: First submitted 2014-05-14; First posted 2014-11-10 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; Dravet syndrome; Seizures; Intractable Epilepsy; Medically Refractory Epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic; Seizures; Drug Resistant Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cannabidiol (Other): open label administration
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol

SUMMARY:
Part A: To evaluate the safety and tolerability of multiple ascending doses of GWP42003-P compared with placebo with respect to:

* Incidence, type and severity of adverse events (AEs)
* Effect on vital signs, including weight
* Effect on 12-lead electrocardiogram (ECG) findings
* Effect on laboratory parameters Part B: To make an assessment of the anti-epileptic efficacy of GWP42003-P compared with placebo with respect to the incidence in convulsive seizures
* To determine the plasma concentration time curves for GWP42003-P and its major human metabolite, following escalating multiple doses of GWP42003-P.
* To investigate the effect of GWP42003-P on the pharmacokinetics of concomitant anti-epileptic drugs (AEDs).
* To evaluate cognitive function, sleep quality and daytime sleepiness, in patients taking GWP42003-P in combination with AEDs.

DETAILED DESCRIPTION:
This multi-center study will consist of two parts: Part A and Part B. Part A will investigate the dose-ranging pharmacokinetics and tolerability of GWP42003-P.

Part B is a 1:1 randomized, placebo-controlled 60 day comparison of GWP42003-P against placebo, at the dose which has been identified by Part A as the maximum tolerated dose. Part B will investigate the efficacy and safety of GWP42003-P.

Following completion of Part B, all patients will be invited to continue to receive GWP42003-P in an open label extension study (which is separate to this protocol).

Part A Following establishment of initial eligibility and baseline measurements, patients will enter Part A at Visit 1 and will begin the two month baseline observation period. Patients will record their number of convulsive seizures, and of other seizures, using an IVRS telephone diary system (recorded twice each day). Each call will take approximately five minutes to complete. Patients will return to the clinic at Visit 2 and the investigator will assess the patient's daily number of convulsive seizures from the patient's IVRS data. Patients who have experienced at least four convulsive seizures (tonic-clonic seizures and/or drop attacks) per month for each of the previous two months) and who meet all of the other inclusion/ exclusion criteria will be eligible to continue in the study. Patients will be asked for information regarding AEs, concomitant medications and/or changes to their medication.

Eligible patients will enter into the pharmacokinetics part of the study at Visit 2 where blood samples will be taken using a sparse sampling strategy to minimize the blood volumes required for analysis of the plasma concentration/time curve for concomitant AEDs and routine safety bloods. This is conducted prior to the administration of Study medication at Dose Level 1.

In each dose level, patients will be randomly assigned so that eight patients receive GWP42003-P and two patients receive placebo in each group. Patients will receive their study medication each day for the seven day exposure period. During this part of the study, patients will continue to record their daily number of convulsive seizures and of other seizures, using an IVRS telephone diary system.

At Day 7 (Visit 3), blood will be taken for analysis of both the plasma concentration/time curve of GWP42003-P and its major metabolite, concomitant anti-epileptic medications and for routine safety purposes. At the end of the dosing period in Part A of the study patients will continue on placebo until they are ready to enter Part B of the study.

Dose Level 2 will follow the same set of procedures as Dose Level 1, but dosing will not start until an evaluation of the clinical and pharmacokinetic results from Dose Group 1 has been completed. Subsequently Dose Groups 3 and 4 will be subject to the same procedures.

When Dose Group 4 has completed the seven day Dosing Period, and subject to assessment of clinical safety and pharmacokinetics, patients will then be invited to continue into Part B, which is the double blind, randomized, placebo-controlled phase to investigate the efficacy and safety of GWP42003-P. There will be a washout period of at least two weeks between the last dosing day in Part A and randomization in Part B.

Part B Patients, from any of the dosing groups, who have completed will be invited to participate into Part B which is a 1:1 randomized, placebo-controlled 60 day comparison of GWP42003-P against placebo. They will receive the dose which was identified by Part A as the maximum tolerated dose. Part B will investigate the efficacy and safety of GWP42003-P.

During Part B, patients will continue to record their number of convulsive seizures and other seizures, using an IVRS telephone diary system (recorded twice each day). Assessments will also be made of cognitive function, nocturnal sleep quality and daytime sleepiness.

Note: Eligible patients who have not previously participated in Part A, and who wish to participate in Part B will begin the two month baseline observation period to establish a baseline. Patients will follow the same procedures as outlined in Visit 1 (of Part A). Patients will record their number of convulsive seizures (and of other seizures), using an IVRS telephone diary system (recorded twice each day).

Part A: The primary endpoint is the safety and tolerability profile of single and multiple ascending doses of GWP42003-P compared with placebo.

The variables for analysis will be the difference in incidence, type and severity of AEs, vital signs, ECG, laboratory, and physical examination parameters of GWP42003-P compared with placebo.

Part B: The primary endpoint is the number of patients experiencing at least a 50% reduction in the number of convulsive seizures (from baseline) on active treatment compared with placebo.

Part A: Pharmacokinetic:

1. GWP42003-P: The plasma concentration/time curve will be described following multiple doses of GWP42003-P, with the aim being to define

   * Cmax
   * tmax
   * AUC0-∞, AUC0-t
   * t½ The analytes for the pharmacokinetic analysis will be CBD and its major human metabolite 7-OH-CBD.
2. Concomitant AEDs: The plasma concentration/time curve for concomitant AEDs will be described pre-treatment, and then after seven days of treatment with GWP42003-P, using a sparse sampling strategy. As far as possible, the plasma concentration/time relationship pre-treatment will be compared with the results following treatment with GWP42003-P.

Part B: Efficacy:

1. Number and type of non-convulsive seizures
2. Cognitive function
3. Sleep quality
4. Caregiver Global Impression of Change

ELIGIBILITY:
Inclusion Criteria:Patients meeting the following criteria will be considered eligible for this study:

* Documentation of a diagnosis of drug resistant epilepsy as evidenced by failure to control siezures despite appropriate trial of four or more Anti-Epileptic Drugs at therapeutic doses. Documentation must include the diagnosis of epilepsy type or epilepsy syndrome (if possible), as well as the underlying case, when known.
* Between 1-3 baseline anti-epileptic drugs at stable doses for a minimum of 4 weeks prior to enrollment. Vagus nerve stimulator, ketogenic diet and modified Atkins diet do not count toward this limit.
* Vagus nerve stimulator must be on stable settings for a minimum of 3 months.
* Written informed consent obtained from the patient or the patient's legal representative must be obtained prior to beginning treatment.

Exclusion Criteria:Exclusion: The patient may not enter the study if ANY of the following apply:

• Treatment with any artisanal preparation containing or possible containing CBD during the month before initiation of the study drug.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Seizure Frequency | Baseline to 1 year
  Number of Seizures

SECONDARY OUTCOMES:
Drug Plasma Levels of Cannabidiol | Baseline, 8 weeks, 6 months
  Lab test to check levels of steady cannabidiol use

CONTACTS AND LOCATIONS:
Overall Officials: Francis Filloux, MD, Principal Investigator — University of Utah; Mathew Sweeney, MD, Study Director — University of Utah; Colin VanOrman, MD, Study Director — University of Utah
Locations (1):
- University of Utah School of Medicine, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No